CLINICAL TRIAL: NCT06996431
Title: Development and Effectiveness of an Innovative Care Model Integrating Mobile Health Support to Promote Weight Management in Adults With Overweight or Obesity: A Stepped-wedge Cluster Randomized Controlled Trial
Brief Title: An Innovative Care Model Integrating Mobile Health Support to Promote Weight Management in Adults With Overweight or Obesity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: WM
Record Dates: First submitted 2025-04-17; First posted 2025-05-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Overweight or Obesity; Physical Activities; Healthy Diet; Weight Change; Body Fat; Muscle Mass
Keywords: ecological momentary assessment; weight management; mHealth; primary care; stepped-wedge; cluster RCT; risk stratification; nurse-led
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized controlled trial will be conducted. This design is considered a type of unidirectional crossover randomized controlled trial (RCT). Stepped-wedge trials evaluate the effect of an intervention implemented at the cluster level. In this design, all clusters initially begin in the control condition. Clusters are then randomized into different sequences, which determine the time point at which each cluster transitions from the control condition to the intervention condition. Once a cluster transitions to the intervention, it remains in that condition for the rest of the study. By the final phase, all clusters, including new participants, will be receiving the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group intervention (Active Comparator): Participants in the control group will receive minimal Intervention. They will not be provided with risk-stratified services.
  Interventions: Behavioral: Minimal Intervention
- EMA-based weight management intervention (Experimental): Participants in the intervention group will join an mobile health (mHealth) weight management program integrating ecological momentary assessment (EMA) via a mobile app, post-EMA counseling, and risk-stratiﬁed coaching. This program provides real-time monitoring and personalized feedback to improve diet and physical activity.
  Interventions: Behavioral: EMA-based weight management intervention

INTERVENTIONS:
Behavioral: EMA-based weight management intervention — Participants will complete four 7-day EMA sessions, reporting their diet for 3 days and physical activity for 4 days by completing ﬁve brief daily mobile app surveys (under 2 minutes each), using a 5-digit case number for privacy. The app automatically retrieves Fitbit data-such as step count, moderate-to-vigorous physical activity (MVPA), sedentary behavior, and heart rate- and sends timely reminders if surveys are missed.
  Within one week after the ﬁrst EMA session, participants will attend a nurse- led counseling session using the 5A Model (Assess, Advise, Agree, Assist, Arrange), providing tailored feedback based on EMA and Fitbit data, and addressing barriers to change. This is followed by risk-based coaching from a dietitian and ﬁtness instructor, with individualized diet and exercise plans. Between sessions, participants receive ongoing support, including instant reminder messaging and weekly motivational messages to encourage healthy behaviors.
  Arms: EMA-based weight management intervention
Behavioral: Minimal Intervention — Participants will not receive risk-stratified services but will be provided with informational leaflets offering general advice on maintaining a healthy diet, regular exercise, smoking cessation, and alcohol cessation.
  Arms: Control group intervention

SUMMARY:
The objective of this clinical trial is to evaluate whether an innovative care model integrating mobile health (mHealth) support improves weight management in adults with overweight or obesity. The primary research questions are: (1) Does the intervention promote weight change at the 6-month follow-up? (2) Does the intervention enhance physical activity and encourage a healthy diet at the 3- and 6-month follow-ups?

To address these questions, researchers will compare the intervention group with a control group to measure changes in weight, physical activity, and dietary habits.

At baseline, all participants will complete a survey assessing demographics, body weight, height, central obesity, lifestyle, weight loss history, and expectations. The intervention group will receive a weight management program based on Ecological Momentary Assessment (EMA), incorporating risk-stratified health services, with follow- ups at 3 and 6 months. The control group will receive minimal intervention in the form of general health advice, with follow-ups at the same intervals.

DETAILED DESCRIPTION:
Background: Obesity leads to cardiovascular diseases, diabetes, musculoskeletal disorders, and many types of cancers. Insufficient physical activity and unhealthy diet (including high intake of saturated fatty acids, fat and inadequate consumption of dietary ﬁbre) are the major causes of obesity but they are preventable and reversible.

The Population Health Survey 2020-22 showed that the overall prevalence of overweight and obese (level 1 and 2) in Hong Kong is 22.0% and 32.6%, respectively. The age-standardized prevalence of physical inactivity has risen from 12.4% (crude prevalence: 13.0%) in 2014-15 to 24.8% in 2020-22. Still 1,486,000 HK residents aged 18 years or above had not met the recommended physical activities level by World Health Organization (WHO). About 4.6% of the population have raised blood glucose or diabetes in 2020-22, compared to 3.9% in 2014-15. The age-standardized prevalence of raised total cholesterol has risen from 38.4% in 2014-15 to 46.5% in 2020-22. About 39.1% of the population eat red meat at least once every day, but only 1.5% of the population intake 2 standard bowls of fruits and 3 bowls of vegetables.

The government targets to reduce a relative 10% of prevalence of physical inactivity by 2025 (compared to 2018) and halt the rise in obesity. The Hong Kong government has been promoting physical activity and healthy diet through public education and social marketing campaigns, but local routine primary healthcare service providers, including Hospital Authority (HA), District Health Centres (DHCs) and non-governmental organizations (NGOs), do not have standard protocols for assessing behavioral risk factors and delivering eﬀective intervention for physical activity and healthy diet.

Mobile Health (mHealth) intervention is a novel and cost-eﬀective approach to increase physical activity, which was highly supported by the WHO. A meta-analysis showed that mHealth intervention was associated with an increase of physical activity at short-(≤ 3 months, by 506 steps per day, 95%CI= -80 to 1092) and long-term (≥6 months, by 753 steps per day, 95%CI= -147 to 1652) follow-up. The meta-analysis also showed that intervention can reduce sedentary time at short-term (≤ 3 months, standardized mean diﬀerences (SMDs)=-0.49, 95%CI= -1.02 to 0.03) follow-up but the result was not statistically signiﬁcant. However, most apps cannot provide personalized intervention and their intervention do not involve behavior change techniques. A qualitative study showed 45.4%of users of smartphone apps disagreed or strongly disagreed that text messages promote them to do more physical activity since those messages did not match their motivation.

To capture the facilitators, barriers, and behaviors in naturalistic settings, ecological momentary assessment (EMA) using mobile devices was developed in recent years. During EMA, users are repeatedly prompted to provide simple information about their experiences and/or behaviors at predetermined and/or random intervals throughout the day. The advantage of EMA includes lower recall bias and providing information at diﬀerent times of the day. Based on EMA summaries, healthcare professionals could design more personalized interventions. EMA information also enables the provision of ecological momentary intervention (EMI), which the software collecting EMA automatically analyze EMA data and provide tailored messages, potentially improving user engagement and compliance to the intervention. EMA and EMI have been adopted in improving mental health, smoking cessation, and reducing substance use with promising results, but interventions for weight management were still under development

Sai Kung, Southern and Wong Tai Sin have set up DHCs or DHC express to deliver health promotion, health assessment, chronic disease screening and educational programs to the residents in these districts. According to the FAMILY Cohort 2011-14, obesity and overweight is the highest reported chronic diseases (Southern: 66.0%; WTS: 63.0%; Sai Kung: 69.0%) in these 3 districts for both male and female. Each DHC has a multidisciplinary healthcare team to oﬀer consultation and health education. As the population ages, there is an increasing demand for intervention, but manpower is limited. Hence a systematic and eﬃcient system in screening, risk stratiﬁcation, and delivering interventions for the overweight is urgently needed. Digital and remote intervention is also valuable to increase DHC clients' uptake of lifestyle intervention as most clients without disease diagnosis normally have lower intention to visit DHC for health coaching. A primary care model with shorter intervention time but suﬃcient human interaction would need to be developed in the DHC setting.

The stepped-wedge cluster randomized controlled trial (SWT) design has become increasingly popular for evaluating interventions implemented at the cluster level. In this design, all clusters start under the control condition. Clusters are randomized into sequences that determine when each cluster transitions to the intervention condition, which continues until the study concludes. In the ﬁnal phase, new participants in all clusters receive the intervention. Compared to individually randomized trials, SWT oﬀers several advantages: (1) reduced within-cluster contamination; (2) lower risk of staﬀ delivering the wrong treatment; (3) increased fairness and acceptance among participants; and (4) reduced resource demands, as clusters are not required to simultaneously prepare for intervention delivery. As a randomized trial, SWT is more robust than quasi-experimental designs. Compared to conventional parallel cluster trials, SWT provides additional beneﬁts: (1) it evaluates interventions across all clusters; (2) facilitates cluster recruitment when intervention eﬀects are promising; (3) accommodates odd or very small numbers of clusters, unlike cluster RCTs that require balanced intervention and control groups; (4) allows for both within-cluster and between-cluster comparisons; and (5) requires fewer clusters to achieve adequate statistical power.

Study design: This study will employ a stepped-wedge cluster randomized controlled trial design. The study period will consist of four consecutive four-month phases. Three non-governmental social service organizations (NGOs) will serve as clusters for randomization. In the ﬁrst phase, all participants across the three clusters will be allocated to the control group. In the second phase, newly recruited participants in Cluster 1, determined randomly, will receive the intervention, while the other two clusters remain in the control group. In the third phase, newly recruited participants in Clusters 1 and 2 will receive the intervention, while Cluster 3 remains in the control condition. In the fourth phase, all newly recruited participants across the three clusters will be allocated to the intervention condition. A web-based portal system will be developed to assist NGO staﬀ in delivering the weight management intervention. During the study, NGO staﬀ will undergo capacity training on study procedures, risk assessment, and using the web-based portal system.

Procedure: Recruitment will be conducted both oﬄine (e.g., posters) and online (e.g., Facebook and Instagram). Interested participants will complete an online form to determine eligibility. Subsequently, recruitment staﬀ (e.g., nurses, ﬁtness instructors, dietitians, or social workers) will contact eligible participants to invite them to an in-person enrollment session. During this session, participants will be briefed about the study, provide informed consent, and undergo baseline health assessments, including anthropometric measurements (e.g., height, weight, waist circumference), body composition analysis (e.g., body fat and muscle mass using the Tanita MC-580 Dual Frequency Segmental Body Composition Analyzer), and self-reported physical activity levels. An optional 5cc blood sample collection will be oﬀered if prior lipid and glucose proﬁles are outdated by more than 28 days, with all samples destroyed after the study. Participants will also complete the Physical Activity Readiness Questionnaire (PAR-Q) and the American College of Sports Medicine (ACSM) Risk Stratiﬁcation Screening Questionnaire to determine their appropriate exercise intensity.

The project coordinator will provide biweekly updates on the number of screenings and enrolled participants. Recruitment eﬃciency will be reviewed and discussed in biweekly and monthly team meetings to identify and implement improvements in recruitment strategies. The three NGOs will be randomly assigned to clusters 1, 2, or 3 using computerized randomization, which will take place one month before recruitment begins. This timeline will allow suﬃcient time to complete staﬀ training. While healthcare workers and participants will not be blinded to their group allocation, data analysts will remain blinded to minimize potential bias during data analysis. Once randomized, participants will remain in their assigned treatment group throughout the study. Any deviations from the protocol will be documented, along with explanations, in future reports.

Intervention Group:

Participants in the intervention group will engage in an mHealth weight management program comprising multiple components: ecological momentary assessment (EMA) using a mobile app, wearable activity tracking, counseling sessions, and risk-based coaching.

Participants will complete four EMA sessions, each lasting 7 days. During these sessions, they will report their diet for 3 days and physical activity for 4 days, completing ﬁve brief daily surveys (under 2 minutes each) via a mobile app developed for both iOS and Android platforms. To protect privacy, participants will use a 5-digit case number instead of personal information. The app will retrieve data from Fitbit devices (e.g., step count, moderate-to-vigorous physical activity, sedentary behavior, heart rate) and prompt participants to complete surveys spaced approximately 4 hours apart. If participants miss a prompt, they will have a 30-minute window to respond, with reminders sent 15 and 5 minutes before the deadline. On 3 selected days, participants will document their food intake using text, audio recognition, and photos.

Participants will utilize Fitbit devices to monitor various physical activity metrics, including step count, moderate-to-vigorous physical activity (MVPA), sedentary behavior, and physiological data such as heart rate and heart rate variability. To complement Fitbit data, participants will also install tracking apps such as Google Fit (for Android) or Apple Health (for iOS) to ensure comprehensive monitoring.

Within one week of completing the ﬁrst EMA session, participants will attend a counseling session delivered by nurses using the 5A model (Assess, Advise, Agree, Assist, Arrange). This session will provide tailored feedback based on EMA data and address barriers to behavior change.

Following this, risk-based coaching will be conducted by a dietitian and ﬁtness instructor, who will provide individualized dietary and physical activity plans, including targeted meal recommendations and home-based exercise programs.

After the ﬁrst EMA session and counseling, participants will proceed to the second EMA session, during which they will receive additional support via instant messaging. The third EMA session will occur one week before the 3-month follow-up, and the fourth EMA session will take place one week before the 6-month follow-up.

Control Group:

Participants in the control group will receive a brief telephone counseling session following their EMA session. This session will provide basic information on physical activity and diet, referencing resources such as the Centre for Health Protection's guides on diet and nutrition and physical activity. After the 6-month follow-up, control group participants will receive the same intervention as the intervention group to ensure equitable access to the program.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥18 years;
2. able to read and communicate in Chinese;
3. own a smartphone with internet access;
4. have good mobility alone without gait aid;
5. body mass index ≥ 23.0;
6. and no contraindication for physical activity as evidenced by: If aged < 70: do not meet any criteria in PAR-Q, or sign declaration of having medical clearance if meet any criteria in PAR-Q; If aged ≥ 70: sign the declaration about conducting physical activity frequently or having medical clearance

Exclusion Criteria:

1. Have a terminal illness (e.g., advanced cancer, dementia, pulmonary, neurological, motor-neuron, and advanced cardiovascular disease) or with a life expectancy of less than 6 months;
2. currently receiving treatment for any cancer (active cancer patients) or cancer survivor of any GI cancers (e.g. colorectal cancer, stomach cancer);
3. lactating, pregnant or planning for pregnancy in the coming 6 months;
4. have current diagnosis of psychiatric disorder;
5. have previous diagnosis of eating disorder;
6. have diagnoses of gastrointestinal conditions (e.g. Irritable Bowel Syndrome, Ulcerative Colitis, Crohn's Disease, Coeliac Disease);
7. currently receiving intensive diet or exercise treatment;
8. have clinical obesity (e.g. confirmation of excess body fat plus limitations of day-to-day activities or signs or symptoms of obesity-related organ dysfunction). Examples of obesity-related organ dysfunction include NAFLD with hepatic fibrosis, the cluster of hyperglycaemia, high triglyceride levels, and low HDL cholesterol levels. Examples of limitations of day-to-day activities include significant age-adjusted limitations of mobility and/or other basic ADL (e.g. bathing, dressing, toileting, continence, eating).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 6-month from baseline
  Defined as the change in weight of participants over a speciﬁed period, this measurement compares the weight change between the intervention and control groups. Participants' weights will be recorded in kilograms at baseline and at a 6-month follow-up using a calibrated digital scale.

SECONDARY OUTCOMES:
Change in weight | 3- and 12-month from baseline
  Defined as the change in weight of participants over a speciﬁed period, this measurement compares the weight change between the intervention and control groups. Participants' weights were recorded in kilograms at baseline, 3- and at a 12-month follow-up using a calibrated digital scale.
Proportion of overweight or obesity | 3-, 6- and 12-month follow-up from baseline
  Deﬁ ned as the percentage of participants classiﬁed as overweight or obese based on their Body Mass Index (BMI). According to the classiﬁcation for Chinese adults in Hong Kong,BMI ≥ 23 kg/m² is defined as overweight, and BMI ≥ 25 kg/m² is defined as obesity. BMI is calculated as a person's weight in kilograms divided by the square of his height in meters (kg/m2).
Proportion of participants with ≥5% weight change | 3-, 6- and 12-month follow-up from baseline
  Defined as the proportion of participants experiencing a weight change of 5% or more from their baseline weight. Weight measurements will be taken in kilograms using a calibrated digital scale at baseline, and at 3-, 6-, and 12-month follow-ups. The proportion will be reported as a percentage (0% to 100%), where higher percentages indicate a greater number of participants with a weight change of 5% or more.
Change in body fat | 3- and 6-month follow-up from baseline
  Deﬁned as the change in body fat mass from baseline to the end of the study period. Body fat mass will be measured in kilograms using the Tanita MC-580 Dual Frequency Segmental Body Composition Analyzer, a body composition analyzer. The scale provides a numeric value for muscle mass. A higher or lower muscle mass indicates a change relative to baseline, with no value inherently representing a better or worse outcome.
Change in muscle mass | 3- and 6-month follow-up from baseline
  Defined as the change in muscle mass from baseline to the specified follow-up periods. Muscle mass will be measured in kilograms using the Tanita MC-580 Dual Frequency Segmental Body Composition Analyzer, a body composition analyzer. The scale provides a numeric value for muscle mass. A higher or lower muscle mass indicates a change relative to baseline, with no value inherently representing a better or worse outcome.
Change in waist circumference | 3-, 6-, and 12-month follow-up from baseline
  Defined as the change in waist circumference from baseline to the specified follow-up periods. Waist circumference will be measured in centimeters using a standard measuring tape. The scale provides a numeric value for waist circumference, with no predetermined minimum or maximum value. An increase or decrease in waist circumference indicates a change relative to baseline, with no value inherently representing a better or worse outcome.
Change in waist-to-hip ratio | 3-, 6-, & 12-month follow-up from baseline
  Defined as the change in the waist-to-hip ratio (WHR) from baseline to the specified follow-up periods. The waist-to-hip ratio will be calculated by dividing the waist circumference (measured at the narrowest point of the torso) by the hip circumference (measured at the widest point of the hips). Both measurements will be taken in centimeters using a standard measuring tape.
Change in self-report time of physical inactivity | 3- and 6-month follow-up from baseline
  Defined as the change in self-reported time spent inactive from baseline to the specified follow-up periods. Physical inactivity is defined by the World Health Organization (WHO) as engaging in less than 150 minutes of moderate- or vigorous-intensity physical activity per week (or an equivalent amount) for persons aged 18 years or older.
  This outcome will be measured using the Global Physical Activity Questionnaire (GPAQ), Chinese version, which assesses physical activity in multiple domains (work, transport, and recreation). The GPAQ provides total physical activity time in minutes per week, with no strict minimum or maximum value.
  Higher scores on the GPAQ reflect more time spent active, while lower scores indicate less time spent active.
Change in self-report time of moderate to vigorous physical activities (MVPA) | 3- and 6-month follow-up from baseline
  Defined as the change in self-reported time spent on MVPA from baseline to the specified follow-up periods. This data will be collected using the Global Physical Activity Questionnaire (GPAQ), Chinese version, which assesses physical activity in multiple domains (work, transport, and recreation).
  The GPAQ calculates the total time spent on MVPA in minutes per week. There is no strict minimum or maximum value for the reported time. Higher scores reflect more time spent on MVPA, while lower scores indicate less time. Changes will be evaluated relative to baseline, with no value inherently representing a better or worse outcome.
Change in diet consumption | 3- and 6-month follow-up from baseline
  Defined as the change in dietary intake from baseline to the specified follow-up periods. Dietary intake includes total calorie consumption and nutrients such as saturated fat, trans fat, carbohydrates, protein, sodium, sugar, and dietary fiber. Data will be collected using 3-day food intake records completed during the first Ecological Momentary Assessment (EMA), the week before the 3-month follow-up, and the week before the 6-month follow-up.
  Participants with extreme underreporting or overreporting of calorie intake, defined as the lowest and highest 1% of reported values, will be excluded from the analysis. Dietary intake values will be presented in standard units (e.g., calories, grams, or milligrams). Higher or lower values for specific nutrients or calorie intake indicate a change relative to baseline.
Dietary adherence to government guideline | 3- and 6-month follow-up from baseline
  Dietary adherence will be assessed based on the Hong Kong Department of Health guidelines for age-adjusted intake of grains, vegetables, fruits, meat, fish, eggs and alternatives, as well as milk and alternatives. Data will be collected at baseline, the 3-month follow-up, and the 6-month follow-up. Adherence will be evaluated using a scoring system, with 1 mark awarded for meeting the recommended intake in each of the 5 dietary components. The maximum total score is 5. The scoring criteria are as follows:
  1. Grains: Male: 4 - 8 bowls; Female: 3 - 6 bowls; Elderly: 3 - 5 bowls
  2. Vegetables: at least 3 servings
  3. Fruits: at least 2 servings
  4. Meat, fish, egg and alternatives: Male: 5 - 8 taels; Female: 5 - 7 taels; Elderly: 5 - 6 taels
  5. Milk and alternatives: Male: 2 glasses; Female: 1 - 2 glasses; Elderly: 1 - 2 glasses
Change in daily step counts | 3- and 6-month follow-up from baseline
  Defined as the change in daily step counts from the first EMA to the 3- and 6-month follow-ups. Step counts will be documented using a step count app and retrieved through the EMA app, providing a daily total of steps.
  Step counts are presented as numeric values, with no predetermined minimum or maximum. A higher or lower daily step count indicates a change relative to baseline, with no value inherently representing a better or worse outcome.
Change in lipid profile | 6-month follow-up from baseline
  Defined as the change in lipid profile from baseline to the 3-month follow-up. The lipid profile will include total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides.
  Lipid levels will be measured in milligrams per deciliter (mg/dL). Changes in lipid profile values will be evaluated relative to baseline, with no specific value inherently representing a better or worse outcome.
Proportion of elevated blood glucose | 6-month follow-up from baseline
  Defined as the proportion of participants with raised blood glucose at baseline and the 3-month follow-up. This is calculated by dividing the number of participants with raised blood glucose by the total number of participants who underwent a blood test.
  Raised blood glucose is defined according to the World Health Organization (WHO) criteria as a fasting plasma glucose concentration ≥ 7.0 mmol/L (126 mg/dL) or being on medication for raised blood glucose. Changes in the proportion will be evaluated relative to baseline.
EMA compliance | baseline
  Defined as the proportion of completed EMA out of all EMA prompts.
Compliance to the counselling | Day 15
  Defined as proportion of attending the counselling after the 1st EMA
Perception and attitude toward the project | 6-month follow-up
  Qualitative feedback on perceptions and attitudes toward the weight management project among participants and NGO staff will be collected using semi-structured interviews. At least 10 participants (5 from each group) and 6 staff members will be interviewed. The interviews will last approximately 30 to 45 minutes.
  The final sample size will depend on data saturation, where no new themes emerge during analysis. Individual interviews will be audio-recorded and transcribed verbatim. Data will be analyzed using thematic analysis to identify key themes and patterns in perceptions and attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Chee Chan Professor, Principal Investigator — he University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Aberdeen Kaifong Welfare Association, Hong Kong
  - Haven of Hope Christian Service, Hong Kong
  - Hong Kong Sheng Kung Hui Welfare Council, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be shared at 2 years after article publication with no end date.
Supporting Information: Study Protocol, ICF